CLINICAL TRIAL: NCT03366324
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of the Combination of Anti-CD19 Chimeric Antigen Receptor-Modified T Cell (CAR-T) Therapy and Hematological Stem Cell Transplantation (HSCT) for MRD+ B-cell Malignancies
Brief Title: Anti-CD19 CAR-T Therapy Combine With HSCT to Treat MRD+ B-cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Sian Medical Technology Co., Ltd (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); The First People's Hospital of Yuhang District (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-CD19-03
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Acute Lymphoblastic Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: The only one group of patients will receive the combination of CAR-T therapy and HSCT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of CAR-T therapy and HSCT (Experimental): After patients achieve MRD- remissions through Second generation CAR-T cells, they will subsequently receive hematological stem cell transplantations within 30 days.
  Interventions: Genetic: Second generation CAR-T cells; Procedure: Hematological stem cell transplantation

INTERVENTIONS:
Genetic: Second generation CAR-T cells — Patients receive CD19 CAR-T cells transduced with a lentiviral vector on days 0, 1, and 2.
Procedure: Hematological stem cell transplantation — Patients receive hematological stem cell transplantations within 3 months after they achieve MRD- remissions after CAR-T therapies.

SUMMARY:
For micro residual disease (MRD) positive patients who have undergone at least 2 cycles chemotherapies for their CD19+ B-cell malignancies, there would be much more risks for them to receive hematological stem cell transplantation (HSCT) than MRD- patients. In order to reduce HSCT-related adverse events for these kind of patients, investigators plan to conduct CAR-T therapies on them first to make them achieve MRD- statuses, and then transfer them to HSCT.

DETAILED DESCRIPTION:
In order to improve prognoses for MRD+ patients who have undergone at least 2 cycles chemotherapies, patients will receive CAR-T therapy before HSCT, once they achieve MRD- remissions, they will subsequently receive HSCT if there are no contraindications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is pathologically and histologically confirmed as CD19 + B cell tumors, and has no effective treatment options currently, such as chemotherapy or autologous hematopoietic stem cell transplantation (auto-HSCT); or patients voluntarily choose CD19 CAR-T cells as a first treatment;
2. The patient is MRD+ (<10%) after at least two cycles of chemotherapies.
3. B cell hematological malignancies include the following three categories:

   * B-cell acute lymphocytic leukemia (B-ALL);
   * Indolent B-cell lymphoma (CLL, FL, MZL, LPL);
   * Aggressive B-cell lymphoma (DLBCL, BL, MCL);
4. < 70 years old;
5. Expected survival time > 6 months;
6. Female patients around childbearing age, negative pregnancy test before trial, and agreed to take effective contraceptive measures during the trial until the last visit;
7. Voluntarily participate in this experiment and sign informed consent by themselves, or legally authorized representative.

Exclusion Criteria:

1. With a history of allo-HSCT;
2. With a history of epilepsy or other central nervous system diseases;
3. The presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within recent six months, or heart disease with cardiac function in any grade 3 (moderate) or 4 ( severe) (according to the New York Heart Association (NYHA) Functional Classification System);
4. Pregnant or lactating women (safety of this therapy for the unborn child is unknown);
5. Not curable active infection;
6. Patients with active hepatitis B or hepatitis C virus infection;
7. Combined use of systemic steroids within two weeks (except use of inhaled steroid recently or currently);
8. Using product of gene therapy before;
9. Creatinine> 2.5 mg / dl (221.0 umol/L); ALT / AST> 3 X the normal amount; Bilirubin> 2.0 mg / dl (34.2 umol/L);
10. Patients suffering from other uncontrolled diseases, and researchers believe that the patient is not suitable for trial;
11. Patients with HIV-infection;
12. Any situation that may increase the risk of patients or interfere with test results.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 200 days from enrollment
  defined as >= Grade 3（NCI CTCAE version 4.03） signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Number of participants with an MRD negative complete remission after CAR-T therapy and HSCT | 2 years from enrollment
  the efficacy of the combination of CAR-T therapy and HSCT will be estimated based on the number of participants who have an MRD negative (flow cytometry) bone marrow aspirate following the treatment

CONTACTS AND LOCATIONS:
Overall Officials: YU HU, M.D., Ph.D, Principal Investigator — Institute of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Institute of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided